CLINICAL TRIAL: NCT03310047
Title: Intra-individual Reproducibility in Nerve Block Duration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Mikkel Herold Madsen, Principal investigator, Nordsjaellands Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Re_Injection
Record Dates: First submitted 2017-10-07; First posted 2017-10-16 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Anesthesia, Regional
MeSH Terms: interventions — Lidocaine; Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: We will use a two-armed crossover design.
  1. Day one; Right side low dose nerve block and left side high dose nerve block
     * Repeated after 24 hours Day three; Left side low dose nerve block and right side high dose nerve block
     * Repeated after 24 hours
  2. Day one; Left side low dose nerve block and right side high dose nerve block
     * Repeated after 24 hours Day three; Right side low dose nerve block and left side high dose nerve block
     * Repeated after 24 hours
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The process of intervention-implementation and intervention will not be in the participant's line of sight.
  Investigators will not be in the room during the intervention. Outcome assessors will not be in the room during the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Right-low, left-high (Experimental): The right-side perineural catheter will be subject to intervention drug Infusion, Lidocaine, 0.5%, 5 mL Lidocaine and the left side perineural catheter will be subject to intervention Infusion, Lidocaine, 0.5%, 10 mL.
  This will be repeated after 24 hours.
  Interventions: Drug: Infusion, Lidocaine, 0.5%, 5 mL; Drug: Infusion, Lidocaine, 0.5%, 10 mL
- Right-high, left-low (Experimental): The right-side perineural catheter will be subject to intervention drug Infusion, Lidocaine, 0.5%, 10 mL Lidocaine and the left side perineural catheter will be subject to intervention Infusion, Lidocaine, 0.5%, 5 mL.
  This will be repeated after 24 hours.
  Interventions: Drug: Infusion, Lidocaine, 0.5%, 5 mL; Drug: Infusion, Lidocaine, 0.5%, 10 mL

INTERVENTIONS:
Drug: Infusion, Lidocaine, 0.5%, 5 mL — A catheter-based perineural infusion of 5 mL Lidocaine 0.5%
  Other Names: Low dose
Drug: Infusion, Lidocaine, 0.5%, 10 mL — A catheter-based perineural infusion of 10 mL Lidocaine 0.5%
  Other Names: High dose

SUMMARY:
An interventional randomized controlled crossover trial, to illuminate if durations in nerve block durations are predictable within the same subject.

DETAILED DESCRIPTION:
An interventional randomized controlled crossover trial, with the purpose to elucidate the reproducibility in nerve block duration on 20 healthy volunteers in Denmark.

There will be two trial arms:

1: Day one; Right side low dose nerve block and left side high dose nerve block. Repeated after 24 hours. Day three; Left side low dose nerve block and right side high dose nerve block. Repeated after 24 hours

2: Day one; Left side low dose nerve block and right side high dose nerve block Repeated after 24 hours Day three; Right side low dose nerve block and left side high dose nerve block Repeated after 24 hours

All volunteers will receive two peripheral nerve blocking catheters adjacent to the common peroneal nerve and will be treated two times on each side with Lidocaine 0.5% 5 mL and 10 mL.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years
2. ASA classification ≤ II

Exclusion Criteria:

1. Allergy to local anaesthetics
2. Body weight 40 kg
3. Possible peripheral nerve injury or disease, including polyneuropathy and diabetes
4. Enrolment or recent participation in studies that may interfere with this study
5. Habitual use of any kind of analgesic medications
6. Anatomic abnormalities preventing successful US-guided Certa Catheter™ insertion.
7. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Duration of insensitivity towards cold | Up to 10 hours
  Time from nerve block onset time (T1) to nerve block remission (T2)

SECONDARY OUTCOMES:
Onset time | Up to 30 minutes
  Time from infusion (T0) to onset (T1) of the nerve blocking effect
Degree of sensory nerve block | Up to 10 hours
  A four step grading-scale of sensory nerve block intensity. 1 = normal, 2 = different, 3 = warm, 4 = no feeling.
Degree of motor nerve block | Up to 10 hours
  A three step grading-scale of motor nerve block intensity. 1 = normal, 2 = decreased strength, 3 = no strength.

CONTACTS AND LOCATIONS:
Overall Officials: Kai L Lange, MD, DMSci, Study Director — Nordsjaellands Hospital
Locations (1):
- Research Unit, Department of Anaesthesiology, Nordsjaellands Hospital Hilleroed, Hillerød, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No